CLINICAL TRIAL: NCT05752123
Title: A Single Site, Open Label Study to Evaluate the Safety and Efficacy of ET-01 Transplantation in Subjects with Transfusion Dependent Β-Thalassemia
Brief Title: A Study to Evaluate the Safety and Efficacy of ET-01 Transplantation in Subjects with Transfusion Dependent Β-Thalassaemia.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Development plan change
Sponsor: EdiGene (GuangZhou) Inc. (Industry)
Collaborators: The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDI-001-002
Record Dates: First submitted 2023-02-16; First posted 2023-03-02 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Transfusion Dependent Beta-Thalassaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ET-01 (Experimental): BCL11A Enhancer modified Autologous Hematopoietic Stem Cells
  Interventions: Biological: ET-01

INTERVENTIONS:
Biological: ET-01 — Recruited participants will receive ET-01 IV infusion after conditioning.

SUMMARY:
This is an open label, single site study to evaluate the safety and Efficacy of ET-01 Transplantation in subjects with Transfusion Dependent β-Thalassaemia.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject and/or subject's legal personal representative fully understand and voluntarily sign informed consent forms;
* 6~35 years old, all gender;
* Diagnosis of transfusion dependent β-thalassemia (β-TDT) as defined by protocol;
* Eligible for autologous stem cell transplant;
* Organs in good function.

Other protocol defined Inclusion criteria may apply.

Key Exclusion Criteria:

* Subjects with associated α-thalassemia;
* Active bacterial, virus, fungal or parasitic infection, including HIV infection, HbsAg and HBV DNA positive, HCV DNA positive, or Treponema Pallidum infection;
* HLA identical sibling or unrelated donors are available;
* Prior allo-HSCT or gene therapy.

Other protocol defined Exclusion criteria may apply.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs & SAEs identified according to NCI CTCAE 5.0. | From ET-01 infusion to 104 weeks post-transplant
All-cause mortality. | From signing of informed consent to 104 weeks post-transplant
Incidence of transplant-related mortality. | within 100 days post-transplant
Proportion of subjects with engraftment. | up to 42 days post-transplant

SECONDARY OUTCOMES:
Change in total hemoglobin from baseline. | within 104 weeks post-transplant
Change of HbF from baseline. | within 104 weeks post-transplant
Change of proportion of HbF/Hb. | within 104 weeks post-transplant
Change of frequency of packed RBC transfusions. | From 6 months before recruitment to 104 weeks post-transplant
Change of volume of packed RBC transfusions. | From 6 months before recruitment to 104 weeks post-transplant

CONTACTS AND LOCATIONS:
Locations (1):
- PLA 923 Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No